CLINICAL TRIAL: NCT05529641
Title: Effects of Combined Diaphragmatic Resistance Training and Cervical Stabilization Exercise in People With Chronic Neck Pain.
Brief Title: Effects of Diaphragmatic Resistance Training in People With Chronic Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, YI-JU TSAI, Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCKU-DRT-2022
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Neck Pain; Diaphragm; Exercise Training; Inhalation
Keywords: Chronic neck pain; Kinematics; Diaphragm; Diaphragmatic resistance training; Stabilization exercise
MeSH Terms: conditions — Neck Pain; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined diaphragmatic resistance training and cervical stabilization exercise group (Experimental): Participants in this group will receive supervised cervical stabilization exercise and diaphragmatic resistance training as home grogram.
  Interventions: Other: Diaphragmatic resistance training; Other: Cervical stabilization exercise
- Cervical stabilization exercise group (Active Comparator): Participants in this group will only receive supervised cervical stabilization exercise.
  Interventions: Other: Cervical stabilization exercise

INTERVENTIONS:
Other: Diaphragmatic resistance training — 6 weeks home exercise of diaphragmatic resistance training will be emphasized.
  Arms: Combined diaphragmatic resistance training and cervical stabilization exercise group
Other: Cervical stabilization exercise — Participants will finish 6 weeks supervised cervical stabilization exercise in person by physical therapist. Dissociated movement and movement control will be emphasized during cervical stabilization exercise.

SUMMARY:
With increasing usage of electronic devices and sedentary lifestyle, chronic neck pain has become a more prevalent musculoskeletal disorder around the world. Many impairments have been identified in people with chronic neck pain including pain, muscle weakness, proprioceptive deficits and altered breathing pattern. Diaphragm is the key muscle for inspiration and also plays an important role in spinal stability. Previous studies have found that diaphragm functions are related to the stability of the lumbar spine through the fascial, neural and visceral systems. Diaphragmatic resistance training thus could have some positive effects on reducing pain and disability in people with low back pain. However, to date how diaphragmatic resistance training would affect chronic neck pain is still unknown. Therefore, the purpose of this study is to investigate the effects of diaphragmatic resistance training on pain, disability and movement quality in people with chronic neck pain.

DETAILED DESCRIPTION:
Chronic neck pain has become a more prevalent musculoskeletal disorder in modern society. The prevalence of chronic neck pain in 2021 gradually increases to 45.7%, that results in a large burden of health care. Chronic neck pain leads to neck motion limitation, motor control impairment and unsmooth motion. In addition, faulty breathing pattern has been identified in 83% of people with chronic neck pain. Diaphragm is the most critical muscle for inspiration and also plays an important role in spinal stability that might relate to spinal instability and pain. Studies have proved that effects of diaphragmatic resistance training on reduce pain and improving quality of life in people with low back pain. Diaphragm connects to the lumbar spine and also to the cervical spine through the fascial, neural and visceral system. However, to our best knowledge, the effects of diaphragmatic resistance training in people with chronic neck pain is still unclear. While many studies have demonstrated that cervical stabilization exercises are able to decrease pain and disability and improve movement quality, the effects of combined diaphragmatic resistance training and cervical stabilization exercise in people with chronic neck pain is still unknown. Therefore, the purpose of this study is to investigate the effects of 6 weeks of diaphragmatic resistance training in combination with cervical stabilization exercises in people with chronic neck pain. Participants with chronic neck pain will be randomly assigned to either (1) combined diaphragmatic resistance training and cervical stabilization exercise group or (2) cervical stabilization exercise group. Each group will receive the same cervical stabilization exercises while group (1) will receive additional diaphragmatic resistance training as home program. All participants will have 2 evaluation sessions at baseline and after 6-week intervention for pain, disability and movement quality.

ELIGIBILITY:
Inclusion Criteria:

* Pain between nuchal line to T1 spinous process lasting over 3 months.

Exclusion Criteria:

* First onset acute neck pain.
* Surgery history.
* Neurological symptoms.
* Respiratory, psychiatric and neuromuscular disorders.
* Smoking, pregnant, cancer.
* Severe anemia or diabetes.
* Core exercise in past 12 months.
* Spine or chest deformity.
* Body mass index (BMI) > 30 kg/m/m.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity using Visual Analog Scale (VAS) | Changes from baseline to 6 weeks when participants finish the intervention.
  Visual Analog Scale (VAS), a self-reported scale, provides 100 mm line that participants will mark the maximal and averaged pain intensity within past 7 days. The length of the line that participants marked would be the intensity of pain. The minimal value will be 0 mm and maximal value will be 100 mm. The longer the length indicates the higher intensity of pain.
Disability using Neck Disability Index (NDI) | Changes from baseline to 6 weeks when participants finish the intervention.
  Neck Disability Index (NDI), a self-reported scale, contains 10 sessions of question to evaluating how severe that functional activity level was affected by neck pain. Each session scores ranging from 0 to 5. Total score range from 0 to 50. The higher the score indicates more disability level.
Cervical kinematics | Changes from baseline to 6 weeks when participants finish the intervention.
  Using optical motion analysis system to assess cervical kinematics for movement quality.
Muscle activation | Changes from baseline to 6 weeks when participants finish the intervention.
  Using surface electromyogram to assess muscle activation pattern.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, National Cheng Kung University, Tainan, Taiwan